CLINICAL TRIAL: NCT05823103
Title: Uterine Septum: Novel Pre-surgical Scoring System to Aid and Standardise Hysteroscopic Metroplasty
Brief Title: New Pre-Surgical Scoring System for Uterine Septum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ebtesama Hospital (Other)
Responsible Party: Principal Investigator, Yehia Shawki, Director of Endoscopy Unit, Ebtesama Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100032023001
Record Dates: First submitted 2023-03-27; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Septate Uterus
Keywords: Hysterscopy; Congenital Uterine Anomaly; Uterine Septum; Septet Uterus; Novel Scoring System; Shawki Septum Scoring System
MeSH Terms: conditions — Septate Uterus; Uterine Anomalies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hysteroscopic Metroplasty using ESHRE ASRM Classification (Active Comparator)
  Interventions: Diagnostic Test: ESHRE ASRM Classification
- Hysteroscopic Metroplasty using Shawki Septum Scoring System (Active Comparator)
  Interventions: Diagnostic Test: Shawki Septum Scoring System

INTERVENTIONS:
Diagnostic Test: Shawki Septum Scoring System — Utilising the novel scoring system to facilitate feasibility and safety of hysteroscopic metroplasty for uterine septum
  Arms: Hysteroscopic Metroplasty using Shawki Septum Scoring System
Diagnostic Test: ESHRE ASRM Classification — Utilising the current classification before performing hysteroscopic metroplasty
  Arms: Hysteroscopic Metroplasty using ESHRE ASRM Classification

SUMMARY:
Comparing surgical outcomes of Hysteroscopic metroplasty for uterine septum when using the standard ESGE or ASRM classifications vs the novel scoring system dubbed Shawki Septum Scoring System.

Outcomes based primarily on completion of the septal correction (no residual parts) and avoiding complications, the most significant of which are uterine perforation.

ELIGIBILITY:
Inclusion Criteria:

* Uterine Septum diagnosed by 3D ultrasound

Exclusion Criteria:

-

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11-18 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Complete Septum Correction | 1 month
  No residual septum on 3D ultrasound
Percentage of patients who had an intra-operative Uterine perforation | during the surgery
  Diminishing the risk of intra-operative perforation of the fundus

CONTACTS AND LOCATIONS:
Overall Officials: Yehia Shawki, MRCOG, Principal Investigator — Endo-Planet
Locations (1):
- Shifa Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 1 year following completion

REFERENCES:
- [Result] Rikken JFW, Kowalik CR, Emanuel MH, Bongers MY, Spinder T, de Kruif JH, Bloemenkamp KWM, Jansen FW, Veersema S, Mulders AGMGJ, Thurkow AL, Hald K, Mohazzab A, Khalaf Y, Clark TJ, Farrugia M, van Vliet HA, Stephenson MS, van der Veen F, van Wely M, Mol BWJ, Goddijn M. The randomised uterine septum transsection trial (TRUST): design and protocol. BMC Womens Health. 2018 Oct 5;18(1):163. doi: 10.1186/s12905-018-0637-6. PMID 30290803
- [Result] Practice Committee of the American Society for Reproductive Medicine. Electronic address: ASRM@asrm.org; Practice Committee of the American Society for Reproductive Medicine. Uterine septum: a guideline. Fertil Steril. 2016 Sep 1;106(3):530-40. doi: 10.1016/j.fertnstert.2016.05.014. Epub 2016 May 25. PMID 27235766
- [Result] Alcazar JL, Carriles I, Cajas MB, Costa S, Fabra S, Cabrero M, Castro E, Tomaizeh A, Laza MV, Monroy A, Martinez I, Aguilar MI, Hernani E, Castellet C, Oliva A, Pascual MA, Guerriero S. Diagnostic Performance of Two-Dimensional Ultrasound, Two-Dimensional Sonohysterography and Three-Dimensional Ultrasound in the Diagnosis of Septate Uterus-A Systematic Review and Meta-Analysis. Diagnostics (Basel). 2023 Feb 20;13(4):807. doi: 10.3390/diagnostics13040807. PMID 36832295
- [Result] Rikken JFW, Kowalik CR, Emanuel MH, Bongers MY, Spinder T, Jansen FW, Mulders AGMGJ, Padmehr R, Clark TJ, van Vliet HA, Stephenson MD, van der Veen F, Mol BWJ, van Wely M, Goddijn M. Septum resection versus expectant management in women with a septate uterus: an international multicentre open-label randomized controlled trial. Hum Reprod. 2021 Apr 20;36(5):1260-1267. doi: 10.1093/humrep/deab037. PMID 33793794
- [Result] Nouri K, Ott J, Huber JC, Fischer EM, Stogbauer L, Tempfer CB. Reproductive outcome after hysteroscopic septoplasty in patients with septate uterus--a retrospective cohort study and systematic review of the literature. Reprod Biol Endocrinol. 2010 May 21;8:52. doi: 10.1186/1477-7827-8-52. PMID 20492650
- [Result] Agostini A, Bretelle F, Cravello L, Ronda I, Roger V, Blanc B. [Complications of operative hysteroscopy]. Presse Med. 2003 May 24;32(18):826-9. French. PMID 12870384